CLINICAL TRIAL: NCT00196209
Title: Randomized Study Comparing Cardioversion vs. Catheter Ablation in Patients With Persistent Atrial Fibrillation
Brief Title: Cardioversion vs. Catheter Ablation for Persistent Atrial Fibrillation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Prof. A. Schömig, Deutsches Herzzentrum Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. C00705
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-03-19 (Estimated); Status verified 2008-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): catheter ablation to treat persistent atrial fibrillation
  Interventions: Procedure: catheter ablation
- 2 (Experimental): cardioversion and drug prophylaxis to treat persistent atrial fibrillation
  Interventions: Procedure: external electric cardioversion

INTERVENTIONS:
Procedure: catheter ablation — catheter ablation to treat persistent atrial fibrillation
  Arms: 1
Procedure: external electric cardioversion — external cardioversion and drug prophylaxis to treat persistent atrial fibrillation
  Arms: 2

SUMMARY:
The aim of this randomized study is to evaluate the efficacy of two different approaches for conversion of persistent atrial fibrillation, the non-invasive one (external electrical cardioversion) and the invasive one (catheter ablation).

DETAILED DESCRIPTION:
This randomized study compares two treatment strategies in patients with persistent atrial fibrillation: Cardioversion vs. catheter ablation. Cardioversion is a low risk standard treatment option for patients with persistent atrial fibrillation. However, mid- and long term efficacy (regarding the maintenance of sinus rhythm) is low. Catheter ablation is an invasive treatment which has been reported to result in up to 60-70% of patients in stable sinus rhythm. However, it is a potentially dangerous invasive procedure with potentially fatal complications.

Comparison: External cardioversion vs. catheter ablation

ELIGIBILITY:
Inclusion Criteria:

* Age >20 years and <75 years
* documented persistent atrial fibrillation for at least 3 months (documented in at least 2 ECGs or holter-ECGs during the previous 3 months before inclusion and persistent atrial fibrillation in a 7-d-holter)
* documented sufficient anticoagulation for at least 4 weeks before inclusion

Exclusion Criteria:

* Paroxysmal atrial fibrillation
* NYHA IV (if recompensation is not possible)
* Contraindication for warfarin
* Disturbance of blood coagulation
* Myocardial infarction, PTCA/stenting, bypass-operation, stroke, intracranial bleeding less than 3 months before
* Reversible causes of atrial fibrillation (i.e. hyperthyroidism)
* Pregnancy
* LA-diameter > 55mm
* LV-function < 30% EF
* Aortic or mitral stenosis or regurgitation III°-IV°
* Prosthetic valves

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2005-08; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Event-free survival after 6 months (i.e. freedom of atrial tachyarrhythmias - as evaluated in a 7-d-holter, stroke, pulmonary vein stenosis - as evaluated in a CT-/MRT-scan 6 months after the initial procedure - and death). | 6 months

SECONDARY OUTCOMES:
success-rate immediately after intervention | success-rate immediately after intervention
need for re-intervention between 2 and 3 months after initial procedure if not stable sinus rhythm at the two-months follow-up (further ablation/cardioversion) | 2-3 months
burden of atrial fibrillation in a 7-day-holter after 6 months | 6 months
significant improvement in exercise capacity (measured by spiroergometry) | 6 months
decrease in NT-pro-BNP levels in the blood after 6 months compared to the level before initial intervention | 6 months
improvement of quality-of-life (combined questionnaire including the SF-36 form) before initial intervention and at the 6-months follow-up | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Deisenhofer, MD, Study Chair — Deutsches Herzzentrum Muenchen; Heidi L Estner, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Germany